CLINICAL TRIAL: NCT05382234
Title: Multisystem Inflammatory Syndrome In Children at Sohag University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Youstena Rashed Attia, Resident docotor pediatric department Facuity Of Medicine Sohag University, Sohag University
Other Study IDs: Soh-Med-22-05-12
Record Dates: First submitted 2022-05-15; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Multisystem Inflammatory Syndrome in Children
MeSH Terms: conditions — pediatric multisystem inflammatory disease, COVID-19 related | interventions — Blood Cell Count

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CBC, ESR ,CRP,Liver Function ,renal function ,ABG,Na,K,D-dimmer ,cardiac enzyme,ferritin ,blood and urine culture in negative cases — cllinical and laboratory evaluation of MIS-C,Effectivness of different therapeutic modalities,Outcome of cases (morbidity,mortality)

SUMMARY:
Since its initial description in December 2019 in Wuhan , China, Corona virus disease 2019 (COVID-19), caused by infection with severe acute respiratory syndrome corona virus 2 (SARS-CoV-2), has rapidly evolved into a worldwide pandemic affecting millions of lives .

Unlike adults, the vast majority of children with COVID-19 have mild symptoms. However, there are children who have significant respiratory disease, and some children may develop a hyper inflammatory response similar to what has been observed in adults with COVID-19. Furthermore, in late April 2020, reports emerged of children with a different clinical syndrome resembling Kawasaki disease (KD) and toxic shock syndrome; these patients frequently had evidence of prior exposure to SARS-CoV-2.

The pathophysiology of MIS-C:

Is unclear ,but it appears to be a consequence of a exacerbated immune system response or maladaptive response of the host .After the virus enters the human cells, the first line of defense against infection should be a quick and well-coordinated immune response ;however, when this mechanism is unregulated and excessive ,hyper inflammation can occur.

Cytokines that play an important role in inducing immunity and immunopathology during infections in excess can cause the clinical syndrome known as cytokine storm. The inflammatory response caused by SARS-CoV-2appears to be the major cause of mortality in infected patients .

The infection of dendritic cells or macrophages by SARS-CoV-2 induces the production of low levels of antiviral cytokines and increases the production of inflammatory cytokines (tumor necrosis factor[TNF], interleukin[IL]-1, IL-6,and interferon ).

ELIGIBILITY:
Inclusion Criteria:

Any suspected case of MIS-C from birth to 12 year included both sexes fulfill criteria of MIS-C (WHO) .

1. Fever for ≥3 days.
2. Clinical signs of multi system involvement (at least 2 of the following):

   1. Rash, bilateral non purulent conjunctivitis, or mucocutaneou inflammation signs (oral, hands, or feet)
   2. Hypotension or shock
   3. Cardiac dysfunction, pericarditis, valvulitis , or coronary abnormalities (including echocardiographic findings or elevated troponin)
   4. Evidence of coagulopathy (prolonged PT or PTT)
   5. Acute gastrointestinal symptoms (diarrhea , vomiting, or abdominal pain)

4. Elevated markers of inflammation (eg ESR, CRP) 5. No other obvious microbial cause of inflammation. 6. Evidence of SARS-CoV-2 infection (Any of the following: Positive SARS-CoV-2 RT-PCR ,positive serology, COVID 19 exposure within the 4 weeks prior to the onset of symptoms).

according to CDC criteria exposure to a patients with suspected or confirmed COVID-19 within the 4 weeks prior to the onset of symptoms.

Exclusion Criteria:

* Other obvious microbial cause of inflammation, including bacterial sepsis and staphylococcal/streptococcal toxic shock syndromes.

Ages: 1 Day to 12 Years | Sex: All
Age Groups: Child
Study Population: Multisystem inflammatory syndrome in children
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Confirmed or suspected cases of Multisystem inflammatory syndrome in children | 1 year
  Confirmed or suspected cases Multisystem inflammatory syndrome in children based On WHO Criteria of MIS-C
  1. Age 0-19 years.
  2. Fever for ≥3 days.
  3. Clinical signs of multi system involvement (at least 2 of the following):
     1. Rash, bilateral non purulent conjunctivitis, or mucocutaneous inflammation signs
     2. Hypotension or shock
     3. Evidence of coagulopathy (prolonged PT or PTT)
     4. Acute gastrointestinal symptoms (diarrhea , vomiting, or abdominal pain)
  4. Elevated markers of inflammation (eg ESR, CRP)
  5. No other obvious microbial cause of inflammation.
  6. Evidence of SARS-CoV-2 infection (Any of the following: Positive SARS-CoV-2 RT-PCR ,positive serology, COVID 19 exposure within the 4 weeks prior to the onset of symptoms).
  according to CDC criteria exposure to a patients with suspected or confirmed COVID-19 within the 4 weeks prior to the onset of symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dong E, Du H, Gardner L. An interactive web-based dashboard to track COVID-19 in real time. Lancet Infect Dis. 2020 May;20(5):533-534. doi: 10.1016/S1473-3099(20)30120-1. Epub 2020 Feb 19. No abstract available. PMID 32087114
- [Background] Riphagen S, Gomez X, Gonzalez-Martinez C, Wilkinson N, Theocharis P. Hyperinflammatory shock in children during COVID-19 pandemic. Lancet. 2020 May 23;395(10237):1607-1608. doi: 10.1016/S0140-6736(20)31094-1. Epub 2020 May 7. No abstract available. PMID 32386565
- [Background] Alunno A, Carubbi F, Rodriguez-Carrio J. Storm, typhoon, cyclone or hurricane in patients with COVID-19? Beware of the same storm that has a different origin. RMD Open. 2020 May;6(1):e001295. doi: 10.1136/rmdopen-2020-001295. PMID 32423970
- [Background] Channappanavar R, Perlman S. Pathogenic human coronavirus infections: causes and consequences of cytokine storm and immunopathology. Semin Immunopathol. 2017 Jul;39(5):529-539. doi: 10.1007/s00281-017-0629-x. Epub 2017 May 2. PMID 28466096